CLINICAL TRIAL: NCT06709365
Title: Tibio-talo-calcaneal Fusion by Hindfoot Nail Versus Open Reduction and Internal Fixation in Treatment of Complex Fractures Distal Tibial and Fragility Ankle Fractures in Elderly
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Abdelgawad Mahmoud, assistant lecturer of orthopaedic surgery, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-24-11-4MD
Record Dates: First submitted 2024-11-25; First posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Fragility Ankle Fractures and Complex Distal Tibial Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fusion group (Active Comparator)
  Interventions: Procedure: Tibiotalar calcaneal fusion by hindfoot
- Open reduction and internal fixation group (Active Comparator)
  Interventions: Procedure: Tibiotalar calcaneal fusion by hindfoot

INTERVENTIONS:
Procedure: Tibiotalar calcaneal fusion by hindfoot — Hindfoot nail for ankle fusion

SUMMARY:
Tibiotalar calcaneal fusion by hindfoot nail Vs open reduction and internal fixation in treatment of complex distal tibial fractures and ankle fragility ankle fractures in elderly

ELIGIBILITY:
Inclusion Criteria:

* pilon fractures complex distal tibial fractures ankle comminuted fractures age more than 65yrs osteoprotic fractures surgically fit patients

Exclusion Criteria:

Ankle fractures unimalleolar undisplaced Pathological fractures Young adults DVT Peripheral vascular diseases Age less than 65 Unfit patient for surgery

-

Ages: 1 Year to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2024-11-30 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
AOFAS American orthopedic foot and ankle score (Score for clinical effects of our intervention) | 2years
  Score for clinical effects of our intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university hospitals, Sohag, Egypt